CLINICAL TRIAL: NCT07173946
Title: Extensive-Stage Small Cell Lung Cancer (ES-SCLC) Prospective, Multicenter, Observational Cohort Study
Brief Title: Prospective Observational Study on ES-SCLC
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K8454
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Extensive-stage Small-cell Lung Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard of Care Anti-tumor Therapy — This is an observational cohort study. There is no intervention assigned by the study protocol. Treatment strategies (including but not limited to chemotherapy, immunotherapy, radiotherapy, and local interventional therapy) are determined solely by the treating physician based on clinical practice guidelines and individual patient circumstances.Patients will receive real-world anti-tumor treatments as prescribed by their physicians. Common treatments for extensive-stage small cell lung cancer (ES-SCLC) may include platinum-etoposide chemotherapy, immune checkpoint inhibitors (such as anti-PD-L1/PD-1 antibodies), radiotherapy, and other therapies per standard clinical practice. The study will observe and record these treatments and their outcomes.

SUMMARY:
Study Title: A Real-World Study on Extensive-Stage Small Cell Lung Cancer (ES-SCLC) What is this study about? This research aims to learn more about how patients with extensive-stage small cell lung cancer (ES-SCLC) are treated in real-world hospital settings and how they respond to those treatments. While new drugs like immunotherapies have shown promise in clinical trials, this study will observe their effectiveness and safety in everyday practice. The goal is to improve future treatment strategies for everyone with this disease.

What will I need to do if I join? This is an observational study. This means your doctors will decide your treatment plan as they normally would. The research team will not assign you any new or experimental treatments.

You will be asked to allow the researchers to collect information from your medical records about your diagnosis, treatment, and health status.

You will need to agree to regular follow-up visits (about every 3 months) by phone or clinic visit so we can track your health over time.

Optional Part: You may choose to provide extra blood and tissue samples (often taken during your routine care) for deeper laboratory research. Scientists will use these samples to try to grow "mini-tumors" (organoids) in the lab to study the disease and test drug responses. You can still participate in the main study even if you decline this part.

What are the benefits? You will receive more structured and consistent follow-up care. If you participate in the optional sample collection, you will receive a 100 RMB subsidy and a personal report on how your mini-tumor reacted to different drugs (this is for informational purposes only and not to guide your treatment).

Your participation will help doctors better understand ES-SCLC and improve care for future patients.

What are the risks or inconveniences? The main inconvenience is the time needed for follow-up visits. If you choose to provide tissue samples, the biopsy procedure itself carries standard risks (like pain, bleeding, or infection), which your doctor will manage carefully.

Your participation is completely voluntary. You can leave the study at any time without giving a reason, and it will not affect your relationship with your doctors or the quality of your medical care.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or above
2. Histologically or cytologically confirmed diagnosis of small cell lung cancer, classified as extensive stage (AJCC 9th Edition Stage IV).
3. Signed informed consent, good compliance, and willingness to undergo treatment and follow-up.
4. Intended to receive any anticancer treatment, including chemotherapy or immunotherapy.

Exclusion Criteria:

1. Lack of definitive histological diagnosis
2. Patients with limited-stage small cell lung cancer
3. Expected survival < 3 months
4. Inability to undergo regular follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age ≥18 years) with histologically or cytologically confirmed extensive-stage small cell lung cancer (ES-SCLC), defined as stage IV according to the AJCC 9th edition cancer staging system, who are scheduled to receive any antitumor therapy (including chemotherapy, immunotherapy, etc.). Participants must provide informed consent and be willing to comply with treatment and follow-up procedures.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of randomization until the date of death from any cause, assessed up to 100 months.
  From date of randomization until the date of death from any cause

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From date of randomization until the date of first documented progression (RECIST v1.1) or death from any cause, whichever occurs first, assessed up to 100 months.
  From the date of randomization to the date of first recording of disease progression ( RECIST v1.1 ) or all-cause death, whichever occurred first.
Objective Response Rate (ORR) | From date of randomization until the date of first documented progression, assessed by RECIST v1.1 criteria at 6- to 8-week intervals up to 100 months.
  From date of randomization until the date of first documented progression, assessed by RECIST v1.1 criteria at 6- to 8-week
Grade ≥3 Adverse Events | From date of first treatment administration until 3 months after last dose, assessed by CTCAE v5.0 criteria.
  The incidence of treatment-related adverse events ≥ grade 3 ( CTCAE v5.0 ).